CLINICAL TRIAL: NCT02882659
Title: Phase I Clinical Trial of Autologous Dendritic Killer Cell-based Immunotherapy for Solid Tumors
Brief Title: Dendritic Killer Cell-based Immunotherapy for Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: FullHope Biomedical Co., Ltd. (Industry)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-07-026B
Record Dates: First submitted 2016-08-18; First posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Colorectal Neoplasms; Hepatocellular Carcinoma; Neoplasm Metastasis
Keywords: Clinical Trial, Phase I
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Hepatocellular; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dendritic Killer Cell (DKC) (Experimental): All enrolled patients received one treatment cycle of DKC cell therapy, which consists of 5 infusion cycles approximately 23 days apart. There were 3 dose levels: 5 x 10^6, 1 x 10^7, and 5 x 10^7 cells, and the protocol followed a traditional 3+3 dose escalation design.
  Interventions: Biological: Dendritic Killer Cell (DKC)

INTERVENTIONS:
Biological: Dendritic Killer Cell (DKC) — DKC is a hybrid cell type capable of dual functionality, i.e. cytotoxicity and antigen presentation, similar to NK cells and DCs, respectively.
  Other Names: FullHope Cell Therapy A (FHCTA)

SUMMARY:
The primary objective of this study is to evaluate the safety of autologous dendritic killer cell (DKC) in patients with metastatic solid tumor and to evaluate the maximum tolerated dose (MTD) of DKC. The primary endpoint of safety evaluation includes physical examination, assessment of vital sign, laboratory test, concomitant medication, and adverse event (AE). The secondary endpoints regarding efficacy includes the generation of tumor specific immune response by detecting CD3+ CD8+ CD69+ IFN-gamma+ T cells, and the improvement of quality of life

ELIGIBILITY:
Inclusion Criteria:

1. Capable and willing of providing signed informed consent before study
2. Patient age ≥20 at date of consent
3. Performance status (ECOG) ≤2
4. Patients have a life expectancy of > 3 months
5. Patients agree to be in compliant to clinical protocol planned treatment plan
6. Histologically confirmed metastatic solid tumor, including colon cancer, gastric cancer, pancreatic cancer, bile duct cancer, liver cancer
7. Patient with histological and conventional imaging proven measurable lesion
8. Patients not pregnant. All male and female patients with reproduction ability should use appropriate contraception method(s) during the study period
9. Patient is not currently under immunosuppressive treatment for previous or recurred autoimmune disease
10. Patient should have received and failed prior standard cancer therapies (according to TVGH standard cancer treatment procedures, or National Comprehensive Cancer Network clinical practice guidelines in oncology)
11. Patient with adequate hematology function:

    Absolute neutrophil count (ANC) ≥ 1,500 cells Total white blood cell (WBC) ≥ 3,000 cells /mm3 Hemoglobin ≥ 9 g/dl Platelets ≥ 100,000 counts /mm3
12. Patient with adequate hepatic and renal function Serum creatinine ≤ 1.5X Upper Limit of Normal (ULN) Total bilirubin (TB) ≤ 1.5X ULN, or ≤ 2.5X ULN for patients with primary HCC or liver metastasis ALT and AST ≤ 2.5X ULN, or ≤ 5X ULN for patients with primary HCC or liver metastasis Alkaline phosphatase (ALP) ≤ 5X ULN
13. Patient showing negative response in syphilis, HIV, HBV and HCV test

Exclusion Criteria:

1. Any other investigational drug used within 28 days prior to first DKC administration
2. Patient with known brain metastasis or metastasis to central nervous system
3. Patient with pulmonary fibrosis
4. Patient with pleural effusion or as cites correspond to CTCAE grading > 2
5. Patient with uncontrolled disease including but not limit to cardiovascular disease, liver disease, renal disease or infectious disease
6. Patients being diagnosed with any cognitive or psychiatric illness
7. Patient not suitable to participate the trial for safety concerns as judged by the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-01 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Safety of DKC as assessed by adverse event (AE) | Entire treatment period (cycle 1-5, 116 +/- 4 days) and follow-up period (452 +/- 4 days)
  The coding system used for AE is MedDRA. Only treatment-emergent adverse events (TEAEs) are considered for primary endpoint. Frequency table of subjects with pre-treatment and treatment-emergent AE are presented by each cohort and overall trial. AE incidents are summarized descriptively by system organ class and preferred term using MedDRA for each cohort and overall trial.
Safety of DKC as assessed by serious adverse event (SAE) | Entire treatment period (cycle 1-5, 116 +/- 4 days) and follow-up period (452 +/- 4 days)
  Serious adverse event incidence is summarized descriptively by system organ class and preferred term for each cohort and overall trial. The causality of SAEs will be assessed by the principal investigator for its relationship to study medication.
Safety of DKC as assessed by dose-limiting toxicity (DLT) | Entire treatment period (cycle 1-5, 116 +/- 4 days) and follow-up period (452 +/- 4 days)
  DLT is defined as Grade ≧ 3 (according to NCI-CTCAE 4.03 grading system), study medication-related (i.e. with causality determined as at least possibly related to study medication), and worsened in comparison to baseline (pre-treatment condition). DLT is determined after first infusion cycle and maximum tolerated dose (MTD) is determined as the highest dose without DLT. DLT is defined by the items listed below:
  Blood and lymphatic system disorders: Grade ≧ 3 of (1) Any febrile neutropenia, (2) Leukocytosis, (3) Anemia
  Other disorders: Grade ≧ 3 of (1) Diarrhea, (2) Vomiting, (3) Fever, (4) Nausea, (5) Anaphylaxis
Safety of DKC as assessed by combining with concomitant anticancer treatment | Entire treatment period (cycle 1-5, 116 +/- 4 days) and follow-up period (452 +/- 4 days)
  The subjects enrolled in the study are cancer patients, who were treated with anticancer drugs before, and possibly during, DKC immunotherapy. Potential adverse drug-drug interaction (DDI) is monitored during treatment and follow-up period.
Safety of DKC as assessed by laboratory examinations | Entire treatment period (cycle 1-5, 116 +/- 4 days) and follow-up period (452 +/- 4 days)
  For each cohort, there are 5 baselines (taken 9 days before infusion) for 5 infusion cycles, and there are 2 evaluation time points in each infusion cycle (at end of first week and second week after infusion) and 4 in the follow-up period (at every 12 weeks). The laboratory evaluation results are tabulated in two aspects: 1) the percentage changes between each evaluation and corresponding baselines, and 2) the mean baseline values of each cycle in each cohort. Laboratory results regarding different functional categories are described separately in following areas.
  Hematology related items: Hb (g/dL), WBC (count/uL), Platelet (x 10^3 count/uL), ANC (count/uL)
  Liver function related items: C-RP (mg/dL), Glucose AC (mg/dL), Total Bilirubin (mg/dL), AST (U/L), ALT (U/L), LDH (U/L), ALP (U/L), gammaGT (U/L)
  Serum lipids and proteins, renal function, and electrolytes related items: HDL-C (mg/dL), Total Cholesterol (mg/dL), Triglyceride (mg/dL), Creatinine (mg/dL), BUN (mg/dL)

SECONDARY OUTCOMES:
Efficacy of DKC as assessed by tumor specific T cell response | Entire treatment period (cycle 1-5, 116 +/- 4 days)
  The tumor specific T cell response was assessed by the detection of CD3+CD8+CD69+IFN-gamma+ T lymphocytes in percentage relative to total peripheral blood mononuclear cells (PBMCs). Baseline value was measured before first infusion cycle, and subsequent evaluation time points were measured right after infusion cycles 2, 3, and 4.
Efficacy of DKC as assessed by change in quality of life | Entire treatment period (cycle 1-5, 116 +/- 4 days) and follow-up period (452 +/- 4 days)
  The quality of life as assessed by the WHO QoL-BREF questionnaire, and the transformed scores (0-100) was used to facilitate the interpretation. Baseline value was measured before first infusion cycle, and evaluation time points were taken right after infusion cycles 2, 3, 4, and 5. During the follow-up period, evaluation time points were taken at every 12 weeks for a total of 4 time points.

CONTACTS AND LOCATIONS:
Overall Officials: Yee Chou, M.D., Ph.D., Principal Investigator — Taipei Veteran General Hospital, Taiwan R.O.C.

IPD SHARING:
Plan to Share IPD: Undecided